CLINICAL TRIAL: NCT04923802
Title: A Multicenter Prospective Observational Study of Non-small Cell Lung Cancer Patients for Development and Validation of Computational Method for Multi-omics-based Neoantigen Prediction and Biomarkers for Immunotherapy Response Evaluation
Brief Title: Multi-Omics Testing for Immunotherapy Efficacy Evaluation (MOTIVATION)
Acronym: MOTIVATION
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit sufficient numbers of patients
Sponsor: GeneCast Biotechnology Co., Ltd. (Industry)
Collaborators: Xinqiao Hospital of Chongqing (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Chest Hospital (Other); Wuhan University (Other); Renmin Hospital of Wuhan University (Other); Tongji Hospital (Other); Southwest Hospital, China (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); People's Hospital of Chongqing (Other); Sichuan Cancer Hospital and Research Institute (Other); The Second Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Guizhou Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shanxi Provincial Cancer Hospital (Unknown); First Hospital of China Medical University (Other); Fujian Provincial Hospital (Other); Peking University Shenzhen Hospital (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: MOTIVATION
Record Dates: First submitted 2021-06-05; First posted 2021-06-11 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer; Neoantigen; Next-generation Sequencing; Biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter prospective observational and exploratory study aims to develop and validate a novel multi-omics-based computational method for neoantigen prediction in non-small cell lung cancer (NSCLC), and discover biomarkers for evaluation of PD-1/PD-L1 inhibitor's efficacy in patients of advanced NSCLC.

DETAILED DESCRIPTION:
Tumor tissues and blood samples from about 400 patients with non-small-cell lung cancer (NSCLC) will be collected for the study, which will be subject to NGS-based genomic, transcriptomic, and methylomic profiling in order to construct a multi-omics landscape of NSCLC. These multi-omics data will be used to construct and validate a novel computational method for neoantigen prediction. Additionally, biomarkers will be explored for prognosis and patient stratification, as well as for evaluation of PD-1/PD-L1 inhibitor treatment efficacy in patients of advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage I-IV non-small cell lung cancer(with no restriction of age, gender, or smoking history)
* Patients in the group will be allowed to collect whole blood and tissue samples at specific time points
* Eastern Cooperative Oncology Group Performance Status of 0-1 within 28 days prior to registration
* No previous systemic anti-tumor therapy
* Signed informed consent

Exclusion Criteria:

* Active or history of autoimmune disease or immune deficiency
* Patients with serious mental disease
* Prior allogeneic stem cell or solid organ transplantation
* Pregnant or lactating women
* Patients who cannot obtain tumor tissue samples and / or whole blood
* Patients with history of blood transfusion within half a year
* Patients with any other malignancy diagnosed within 5 years
* Received systemic anti-tumor therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-IV non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival (PFS) is defined as the period a participant remains alive without disease progression after study registration. Tumor status is assessed per the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) by computed tomography (CT), positron emission tomography (PET) CT and/or X rays.
  Complete Response (CR) = Disappearance of all lesions Partial Response (PR) = ≥30% decrease in the sum of the lesion diameters Overall Response (OR) = CR + PR Progressive disease (PD) = 20% increase in the sum of lesion diameters, and/or the appearance of 1+ new lesion(s) Stable disease (SD) = Small changes that do not meet any of the above criteria
Disease-free survival (DFS) | 2 years
  Disease-free survival (DFS) is defined as the number of participants remaining alive without disease progression (PD), symptomatic deterioration or death due to any cause. DFS is assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, as follows.
  Complete Response (CR) = Disappearance of all target lesions Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions Progressive disease (PD) = 20% increase in the sum of the diameters of target lesions (must be > 5 mm), unequivocal progression of non-target lesions, and/or the appearance of one or more new lesion(s) Stable disease (SD) = Small changes that do not meet any of the above criteria. The outcome will be reported as the number of participants who meet the criteria for DFS, a number without dispersion.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival (OS) defined as the duration from study registration until death due to any cause. The outcome will be reported as the number of participants known to be alive at 24 months after study registration, a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhu, Principal Investigator — Xinqiao Hospital of Chongqing
Locations (1):
- Second Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No